CLINICAL TRIAL: NCT03920670
Title: Comparison of the ToFscan and TetraGraph During Recovery of Neuromuscular Function in the Post Anesthesia Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-011298
Record Dates: First submitted 2019-02-13; First posted 2019-04-19 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-03

CONDITIONS: Residual Neuromuscular Blockade
Keywords: Neuromuscular Blockade; ToFscan; Tetragraph; AMG; EMG
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Tetragraph (TG) (Experimental): TetraGraph placed on dominant hand, ToFscan placed on non-dominant hand
  Interventions: Device: TetraGraph (TG); Device: ToFscan (TS)
- ToFscan (TS) (Active Comparator): ToFscan placed on dominant hand, TetraGraph (TG) placed on non-dominant hand
  Interventions: Device: TetraGraph (TG); Device: ToFscan (TS)

INTERVENTIONS:
Device: TetraGraph (TG) — TetraGraph device is a neuromuscular transmission monitor capable of estimating the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to percutaneous electrical neurostimulation. Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis will be measured.
Device: ToFscan (TS) — ToFscan is a nerve stimulator module used for the measurement of neuromuscular transmission via accelerometry. ToFscan was developed by Drager Technologies, Canada, and it uses a three-dimensional piezoelectric sensor that attaches to the thumb via a hand adapter to measure acceleration in multiple planes (Murphy et al, 2018). Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis will be measured.

SUMMARY:
The aim of this investigation is to compare the performance of two quantitative monitors utilized on post-anesthesia recovering patients. The ToFscan (Draeger Medical Inc., Telford, PA) represents one of the few standalone acceleromyography (AMG)-based quantitative monitors available for routine clinical use in the United States. The TetraGraph (Senzime AB, Uppsala, Sweden) is a standalone electromyography (EMG)-based quantitative monitor that recently received Conformité Européene (CE) approval. While both of these quantitative monitors can be utilized to guide intraoperative NMBA re-dosing and confirm recovery, they provide their objective data via drastically different techniques.

ELIGIBILITY:
Inclusion Criteria

* Age > or = 18 years old
* Patients willing to participate and provide an informed consent
* Patients undergoing an elective surgical procedure that requires use of non-depolarizing NMBA agents administered intraoperatively.

Exclusion Criteria

* Patients with unilateral disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture, or any similar wrist injury.
* Patients with systemic neuromuscular diseases such as myasthenia gravis
* Patients with significant organ dysfunction that can significantly affect pharmacokinetics of neuromuscular blocking and reversal agents, i.e., severe renal impairment or end-stage liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Ross Renew, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
- University of Debrecen, Debrecen, Hungary

REFERENCES:
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear TD, Deshur M, Benson J, Newmark RL, Maher CE. Comparison of the TOFscan and the TOF-Watch SX during Recovery of Neuromuscular Function. Anesthesiology. 2018 Nov;129(5):880-888. doi: 10.1097/ALN.0000000000002400. PMID 30130260
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Tetragraph (TG) Dominant Hand ToFscan (TS) Non-dominant Hand: TetraGraph was placed on dominant hand, ToFscan (TS) was placed on non-dominant hand
  TetraGraph device is a neuromuscular transmission monitor capable of estimating the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to percutaneous electrical neurostimulation. Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
  ToFscan is a nerve stimulator module used for the measurement of neuromuscular transmission via accelerometry. ToFscan was developed by Drager Technologies, Canada, and it uses a three dimensional piezoelectric sensor that attaches to the thumb via a hand adapter to measure acceleration in multiple planes (Murphy et al, 2018). Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
- ToFscan (TS) Dominant Hand TetraGraph (TG) Non-dominant Hand: ToFscan was placed on dominant hand, TetraGraph (TG) was placed on non-dominant hand
  TetraGraph device is a neuromuscular transmission monitor capable of estimating the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to percutaneous electrical neurostimulation. Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
  ToFscan is a nerve stimulator module used for the measurement of neuromuscular transmission via accelerometry. ToFscan was developed by Drager Technologies, Canada, and it uses a three dimensional piezoelectric sensor that attaches to the thumb via a hand adapter to measure acceleration in multiple planes (Murphy et al, 2018). Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
Period: Overall Study
Arm/Group | Tetragraph (TG) Dominant Hand ToFscan (TS) Non-dominant Hand | ToFscan (TS) Dominant Hand TetraGraph (TG) Non-dominant Hand
Started | 60 | 60
Completed | 57 | 58
Not Completed | 3 | 2
Not completed — Protocol Violation | 2 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tetragraph (TG) Dominant Hand ToFscan (TS) Non-dominant Hand: TetraGraph was placed on dominant hand, ToFscan was placed on non-dominant hand
  TetraGraph device is a neuromuscular transmission monitor capable of estimating the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to percutaneous electrical neurostimulation. Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
  ToFscan is a nerve stimulator module used for the measurement of neuromuscular transmission via accelerometry. ToFscan was developed by Drager Technologies, Canada, and it uses a three dimensional piezoelectric sensor that attaches to the thumb via a hand adapter to measure acceleration in multiple planes (Murphy et al, 2018). Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
- Total: Total of all reporting groups
Arm/Group | Tetragraph (TG) Dominant Hand ToFscan (TS) Non-dominant Hand | ToFscan (TS) Dominant Hand TetraGraph (TG) Non-dominant Hand | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (15.2) | 55.6 (15.1) | 55.6 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 24 | 22 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Mean Train-of-Four Ratios (TOFR's)
Description: Train-of-four ratios is the ratio of the fourth muscle response to the first one.
Time Frame: baseline, after 5 minutes, after + 10 minutes
Population: Dominant arm Train-of-Four Ratios collected for analysis
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Tetragraph (TG) Dominant Hand ToFscan (TS) Non-dominant Hand: TetraGraph was placed on dominant hand, ToFscan was placed on non-dominant hand
  TetraGraph device is a neuromuscular transmission monitor capable of estimating the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to percutaneous electrical neurostimulation. Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
  ToFscan is a nerve stimulator module used for the measurement of neuromuscular transmission via accelerometry. ToFscan was developed by Drager Technologies, Canada, and it uses a three dimensional piezoelectric sensor that attaches to the thumb via a hand adapter to measure acceleration in multiple planes (Murphy et al, 2018). Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
  Dominant arm Train-of-Four Ratios collected for analysis
- ToFscan (TS) Dominant Hand TetraGraph (TG) Non-dominant Hand: ToFscan was placed on dominant hand, TetraGraph (TG) was placed on non-dominant hand
  TetraGraph device is a neuromuscular transmission monitor capable of estimating the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to percutaneous electrical neurostimulation. Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
  ToFscan is a nerve stimulator module used for the measurement of neuromuscular transmission via accelerometry. ToFscan was developed by Drager Technologies, Canada, and it uses a three dimensional piezoelectric sensor that attaches to the thumb via a hand adapter to measure acceleration in multiple planes (Murphy et al, 2018). Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
  Dominant arm Train-of-Four Ratios collected for analysis
Arm/Group | Tetragraph (TG) Dominant Hand ToFscan (TS) Non-dominant Hand | ToFscan (TS) Dominant Hand TetraGraph (TG) Non-dominant Hand
Number analyzed (Participants) | 57 | 58
Ratio
  baseline | 0.97 (0.18) | 0.94 (0.13)
  after 5 minutes | 0.96 (0.20) | 0.95 (0.12)
  after + 10 minutes | 0.99 (.014) | 0.94 (0.12)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of scan, for a total of approximately 10 minutes
Groups:
- Tetragraph (TG) Dominant Hand ToFscan (TS) Non-dominant Hand: TetraGraph was placed on dominant hand, ToFscan was placed on non-dominant hand
  TetraGraph (TG): AMG and EMG neuromuscular blockade monitoring. The TetraGraph device is a neuromuscular transmission monitor capable of estimating the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
  ToFscan (TS): Neuromuscular transmission monitor. A measure of muscle relaxation on an anesthetized subjects. Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
- ToFscan (TS) Dominant Hand TetraGraph (TG) Non-dominant Hand: ToFscan was placed on dominant hand, TetraGraph (TG) was placed on non-dominant hand
  TetraGraph (TG): AMG and EMG neuromuscular blockade monitoring. The TetraGraph device is a neuromuscular transmission monitor capable of estimating the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
  ToFscan (TS): Neuromuscular transmission monitor. A measure of muscle relaxation on an anesthetized subjects. Following simultaneous ulnar nerve stimulation on each arm, the response of the adductor pollicis was measured.
Arm/Group | Tetragraph (TG) Dominant Hand ToFscan (TS) Non-dominant Hand | ToFscan (TS) Dominant Hand TetraGraph (TG) Non-dominant Hand
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/115
Other Adverse Events (participants affected / at risk) | 0/115 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT03920670/Prot_SAP_000.pdf